CLINICAL TRIAL: NCT04118296
Title: Decreasing Severity of Acne Vulgaris After the Use of a Combination of Anti-Acne Cream in West Jakarta
Brief Title: Decreasing Severity of Acne Vulgaris After the Use of a Combination of Anti-Acne Cream
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sukma Skin Treatment (Other)
Responsible Party: Principal Investigator, Jessica Elizabeth, Co-Researcher, Sukma Skin Treatment
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SST-02-2019
Record Dates: First submitted 2019-10-03; First posted 2019-10-08 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Intervention Model Description: This research is a clinical trial research with an experimental research design. Epidemiological association analysis is obtained by calculating Relative Risk (RR) because the research use experimental design and the nature of the two variables studied is categorical.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Intervention will be given in the form of the use of anti-acne combination creams that contain active substances such as Clindamycin 3%, Dexamethasone 0.05% and Tretinoin 0.05%
  Interventions: Drug: Anti-Acne Preparations for Topical Use

INTERVENTIONS:
Drug: Anti-Acne Preparations for Topical Use — Combination of anti acne cream that contain active substances such as Clindamycin 3%, Dexamethasone 0.05% and Tretinoin 0.05%

SUMMARY:
This study was conducted to see whether there was a decrease in the degree of acne vulgaris / pimple, to find out what proportion of respondents experienced a decrease in severity and who did not experience a decrease in the severity of acne vulgaris after the use of an anti-acne cream combination containing active ingredients such as; Tretinoin 0.05% (derivatives of Vitamin A), Clindamycin 5% (antibiotics), and Dexamethasone 0.05% (anti-inflammatory) for 1 month of use.

DETAILED DESCRIPTION:
This research was conducted based on the results of epidemiological studies that the group of adolescents aged 14-19 years had a fairly high prevalence of acne vulgaris, which amounted to 83-85% for female, 95-100% for male and this prevalence rate was increasing over the years. Acne vulgaris is not a dangerous disease, but has a large enough impact for sufferers, especially teenagers. Physical and psychological effects can cause anxiety, depression, and reduce the confidence of sufferers.

Many drugs for acne vulgaris are sold freely and can be bought by everyone without the need to consult a doctor first, coupled with the lack of knowledge of adolescent groups about acne vulgaris and its treatment options, this causes the lack of accurate acne treatment and increases the risk of effects side of the drug. The use of topical medicines in the form of a combination of anti-acne cream is one of the best choices because all the components needed to deal with acne can be combined to become one so that it is more effective and efficient

The short-term goal of this research is to find out what proportion of respondents with mild, moderate and severe acne before being given an intervention in the form of using a combination of anti-acne cream, the proportion of respondents with mild, moderate and severe acne after being given an intervention, the proportion of respondents who were given intervention and experienced decrease the severity of acne vulgaris, and find out the relationship between the use of a combination of anti-acne cream with a decrease in the severity of acne vulgaris.

This research is an experimental design clinical trial research. The research hypothesis is that the use of a combination of anti-acne creams can reduce the severity of acne vulgaris. The study population and sample were in the form of a group of adolescents aged 14-19 years, located in the sampling area, and met the inclusion criteria. The number of samples is 186 respondents .

The ingredients contained in the combination of anti-acne creams are commonly used ingredients and are one of the first-line treatments for acne vulgaris, namely Tretinoin 0.05% (Vitamin A derivatives), Clindamycin 3% (antibiotics), and Dexamethasone 0.05% (anti-inflammation). Based on the literature it is known that these three active substances have proven to be effective in treating acne vulgaris. Side effects can occur mild and not like irritation, skin peeling, redness, and local allergic reactions. These side effects can be minimized by using according to doctor's instructions and will disappear if the use of the cream is stopped.

We researchers always uphold the investigator's ethics and professionalism while conducting this research, and do not fight the medical oath we have taken.

ELIGIBILITY:
Inclusion Criteria:

* respondents aged 14-19 years
* suffering from mild, moderate or severe degree of acne vulgaris in the face area regardless of the respondent's skin type
* agreed to informed consent
* agreed to use a combination of anti-acne creams only and stopped all other skin treatments on the face for at least 3 days

Exclusion Criteria:

* respondents with other skin diseases on the face such as atopic dermatitis, contact, rosacea, viral infections, impetigo, fungal infections, acne eruption
* respondents who are suspected of having allergies to active substances contained in a combination of anti-acne creams

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2019-11-06 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Knowing the relationship & possibility between the use of a combination of anti-acne cream with a decrease in the severity of acne vulgaris | The severity of acne vulgaris is measured after 1 month of use of the combination of anti-acne cream
  Epidemiological association analysis is obtained by calculating Relative Risk (RR).
  If RR = 1, it means that the probability of a severe degree of acne vulgaris with a moderate degree of acne vulgaris is the same as the degree of acne reduction.
  If RR> 1, it means that the possibility of severe acne vulgaris group with moderate acne vulgaris is greater for a decrease in acne degree.
  If RR <1, it means that the possibility of severe acne vulgaris group with moderate acne vulgaris is smaller to experience a decrease in acne degree.

CONTACTS AND LOCATIONS:
Locations (1):
- SMKN 35 Jakarta Barat, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No
Because the respondent's personal data is confidential and it's written in the informed consent that the researcher will not share the respondent's personal data

REFERENCES:
- [Result] Perkins AC, Cheng CE, Hillebrand GG, Miyamoto K, Kimball AB. Comparison of the epidemiology of acne vulgaris among Caucasian, Asian, Continental Indian and African American women. J Eur Acad Dermatol Venereol. 2011 Sep;25(9):1054-60. doi: 10.1111/j.1468-3083.2010.03919.x. Epub 2010 Nov 25. PMID 21108671
- [Result] Ray C, Trivedi P, Sharma V. Acne and Its Treatment Lines. International Journal of Research in Pharmaceutical and Biosciences. 2013 January 23; 3(1): p. 1-16
- [Result] Cunliffe W, Gollnick H. Topical Theraphy. In Cunliffe WJ GH. Acne Diagnosis and Management. London: Martin Dunitz Ltd; 2001. p. 107-114.
- [Result] Katsambas A, Dessinioti C. New and emerging treatments in dermatology: acne. Dermatol Ther. 2008 Mar-Apr;21(2):86-95. doi: 10.1111/j.1529-8019.2008.00175.x. PMID 18394082
- [Result] Rathi SK. Acne vulgaris treatment : the current scenario. Indian J Dermatol. 2011 Jan;56(1):7-13. doi: 10.4103/0019-5154.77543. PMID 21572783
- See also: Acne Vulgaris — https://emedicine.medscape.com/article/1069804-overview#a6
- See also: Clindamycin Topical — https://medlineplus.gov/druginfo/meds/a609005.html